CLINICAL TRIAL: NCT04761146
Title: A Safety and Efficacy Study of Intra-tumoural Diffusing Alpha Radiation Emitters (DaRT) for the Treatment of Primary and Recurrent Squamous Cell Carcinoma of the Vulva
Brief Title: A Safety and Efficacy Study of Intra-tumoural Diffusing Alpha Radiation Emitters for the Treatment of Vulva Cancer
Acronym: DaRT-V
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CCTU- Cancer Theme (Other)
Collaborators: Alpha Tau Medical LTD. (Industry)
Responsible Party: Sponsor-Investigator, CCTU- Cancer Theme, Dr Li Tee Tan, Cambridge University Hospitals NHS Foundation Trust
Organization: Cambridge University Hospitals NHS Foundation Trust (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: DaRT-V
Record Dates: First submitted 2021-02-05; First posted 2021-02-18 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Vulva Cancer, Recurrent; Vulvar Squamous Cell Carcinoma; Vulva Cancer
Keywords: Medical Device; Brachytherapy; Diffusing Alpha-emitters
MeSH Terms: conditions — Vulvar Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DaRT Diffusing Alpha-emitters Radiation Therapy (Experimental): DaRT Diffusing Alpha-emitters Radiation Therapy using the DaRT applicator and seeds, inserted for 14 days prior to removal.
  Interventions: Radiation: DaRT Diffusing Alpha-emitters Radiation Therapy

INTERVENTIONS:
Radiation: DaRT Diffusing Alpha-emitters Radiation Therapy — DaRT is a brachytherapy treatment comprising stainless-steel 316LVM wires coated with radium-224 (Alpha DaRT seeds). The radioactive seeds are inserted directly into the tumour on the perineum and will be removed after 14 days.

SUMMARY:
An investigation to investigate the use of diffusing alpha-emitters radiation therapy (DaRT) for the treatment of new and recurrent squamous cell carcinoma of the vulva.

DETAILED DESCRIPTION:
Squamous cell carcinoma of the vulva is a rare cancer accounting for less than 1% of female cancers. The disease predominantly affects women over the age of 65 although the incidence in younger women is rising, a finding that has been attributed to the effect of increasing human papillomavirus (HPV) infection .

The standard treatment for the primary tumour is surgical excision with the aim of achieving a 1 cm clear margin on histopathology. This requires the surgeon to remove 1.5-2 cm of surrounding normal tissue to allow for shrinkage after tissue fixation. Depending on the size and location of the tumour, the surgical procedure could vary from a wide local excision to a radical vulvectomy, including excision of adjacent structures such as the clitoris, lower urethra or anus, and/or reconstructive surgery. Wound infection and breakdown are common short-term complications of radical vulva surgery. Long term consequences include functional, cosmetic, psychological and psychosexual sequelae, which can have a significant negative impact on quality of life.

Recurrence rates for vulva squamous cell carcinomas range from 15% to 33%. Local recurrence in the vulva is the most common site of relapse (70%) with the groin nodes affected in 24%, pelvic nodes in 16% and distant metastases in 19%. The treatment of choice for local recurrence is surgical excision and 5-year survival rates of up to 45% have been reported. However, patients can develop multiple recurrences over a period of time and the feasibility of surgery becomes increasingly more limited as more and more tissue is removed.

Brachytherapy is a form of radiotherapy where radiation sources are placed directly in contact with or into (interstitial) cancerous tissue. The radiation emitted has a short range in tissue and the brachytherapy dose distribution conforms tightly to the location of the sources with minimal dose to the surrounding healthy tissues.

Alpha Tau Medical Ltd. proposes a novel treatment for malignant tumours using intra-tumoural alpha radiation, which is delivered using the Alpha DaRT Device (Alpha DaRT applicator + Alpha DaRT seeds). The technique, known as Diffusing Alpha-emitters Radiation Therapy (DaRT), combines the advantages of conventional interstitial brachytherapy with the destructive power of alpha particles.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed or recurrent (local) vulva cancer with or without distant metastases
* Histopathological confirmation of squamous cell carcinoma
* Macroscopic tumour in situ (i.e. tumour not excised)
* Age 18 years and over
* ECOG performance status 0-2
* Life expectancy more than 6 months
* Willing and able to give written informed consent to participate
* Measurable target according to RECIST v1.1
* Tumour size ≤ 7 centimetres in the longest diameter
* Target is technically amenable for full coverage by the DaRT seeds

Exclusion Criteria:

* Non-squamous histology
* Concomitant illnesses which may increase risk of radiation toxicity e.g. autoimmune diseases, vasculitis, etc.
* Concomitant immunosuppressive and/or long-term corticosteroid treatment
* Involvement in other studies that may affect evaluation of response or toxicity of DaRT in the past 30 days or 5 half-lives of the investigational product, whichever is longer
* Pregnancy or breastfeeding
* Women of child-bearing potential unwilling to use adequate contraception for the duration of the study and 6 months after completion (further details in CIP section 13)
* Nodal recurrence without local recurrence
* Previous diagnosis of other malignancy < 3 years of enrolment (excluding non-melanomatous skin cancer)
* No concurrent chemotherapy
* Patients who have received prior chemotherapy or targeted therapy require a 1-month washout before DaRT insertion
* Requirement to start chemotherapy within 6 weeks of DaRT insertion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligibility based on sex assigned at birth
Enrollment: 10 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Assess the feasibility of DaRT by the safety of DaRT for the treatment of Primary and Recurrent Squamous Cell Carcinoma of the Vulva | 6 months
  Measuring the feasibility of using the device by the treatment-related adverse events in the follow-up period (graded 1 'not significant' to 5 'death' with Common Terminology Criteria for Adverse Events v5.0)

SECONDARY OUTCOMES:
Assess the efficacy of DaRT for the treatment of Primary and Recurrent Squamous Cell Carcinoma of the Vulva | Day 28 (4 weeks)
  Tumour response at 4 weeks (Day 28) after DaRT insertion as assessed by Response Evaluation Criteria in Solid Tumours (RECIST, complete response to progressive disease) criteria
To evaluate the effect DaRT on the immunological response | 4-6 weeks
  Histological evidence of necrosis in pathological lymph nodes if removed.
Assess the efficacy of DaRT for the treatment of Primary and Recurrent Squamous Cell Carcinoma of the Vulva | 6 months
  Local control rate at 3-month and 6-month follow-up visits
Assess the efficacy of DaRT for the treatment of Primary and Recurrent Squamous Cell Carcinoma of the Vulva | 6 months
  Patient numerical rating scale (NRS) pain score, '0' representing "no pain" to '10' representing "extreme pain"
Assess the efficacy of DaRT for the treatment of Primary and Recurrent Squamous Cell Carcinoma of the Vulva | 6 months
  Patient mental state using the European Organisation for Research and Treatment of Cancer Quality of Life questionnaire. Scored 1-4 from 'Not at All' to 'Very Much'
Assess the efficacy of DaRT for the treatment of Primary and Recurrent Squamous Cell Carcinoma of the Vulva | 4-6 weeks
  Percentage of necrotic tissue if residual tumour is removed surgically
Assess the efficacy of DaRT for the treatment of Primary and Recurrent Squamous Cell Carcinoma of the Vulva | 6 months
  Patients physical state using the European Organisation for Research and Treatment of Cancer Quality of Life questionnaire. Scored 1-4 from 'Not at All' to 'Very Much'

CONTACTS AND LOCATIONS:
Overall Officials: Li Tee Tan, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Cambridge University Hospitals NHSFT, Cambridge, Cambridgehire, United Kingdom

IPD SHARING:
Plan to Share IPD: No